CLINICAL TRIAL: NCT06936163
Title: Surgical Outcomes of Foot Deformities in Hereditary Spastic Paraplegia: A Prospective Cohort Study
Brief Title: A Prospective Cohort Study of Surgical Treatment for Foot Deformities in HSP
Acronym: HSP
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Cao, Professor, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-034(K)
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Spastic Paraplegia
Keywords: Hereditary Spastic Paraplegia; foot deformities
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Foot Deformities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HSP patients (ages 10 to 45) with foot deformities unresponsive to conservative therapy: Patients aged 10 to 45 years who have been diagnosed with isolated Achilles tendon contracture or equinovarus cavus deformity due to hereditary spastic paraparesis (HSP) will be recruited for the study. Eligible participants must have undergone standard conservative treatments, including pharmacological therapy or rehabilitation exercises, but have demonstrated a poor response or progressive worsening of gait disturbances and foot deformities, and be capable of walking barefoot for 10 meters, with or without the use of assistive devices.

SUMMARY:
Through a prospective cohort study, we aim to dynamically evaluate the long-term benefits and risks associated with surgical interventions for hereditary spastic paraparesis (HSP) accompanied by foot deformities. Our goal is to systematically summarize clinical experiences to guide practice and ultimately optimize patient outcomes.

The core research objectives include elucidating:

1. the long-term efficacy of foot deformity correction procedures;
2. the optimal timing for surgical intervention;
3. the establishment of objective evaluation criteria to guide therapeutic decision-making.

DETAILED DESCRIPTION:
Hereditary spastic paraplegia (HSP) is a neurodegenerative disorder characterized by axonal degeneration of the corticospinal tract. This degeneration often leads to foot deformities such as equinovarus, cavus foot, and Achilles tendon contracture, which result from lower limb spasticity and muscular imbalance. These deformities result in gait abnormalities, uneven plantar pressure distribution, and secondary osteoarticular damage, which significantly impair motor function and quality of life. Surgical correction serves as the primary intervention to address fixed deformities and delay disease progression.This prospective, open-label, single-center study aims to evaluate the long-term functional outcomes of surgical treatment for HSP-related foot deformities, determine the optimal timing for surgical intervention, and establish objective evaluation criteria. Over a 2-year period, 100 patients aged 10-45 years with HSP-confirmed isolated Achilles tendon contracture or equinovarus cavus foot deformity will be enrolled in the study. Eligible patients must exhibit progressive deformity refractory to conservative therapy, accompanied by walking pain, frequent falls, and significant quality-of-life impairment. They must also retain the ability to walk independently or with assistive devices for at least 10 meters. All participants will undergo regular clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 10 to 45 years old.
2. Clinically and molecular genetically confirmed diagnosis of hereditary spastic paraparesis (HSP) with either isolated Achilles tendon contracture or equinovarus cavus deformity.
3. Radiographic (X-ray) or computed tomography (CT) evidence confirming the presence of isolated Achilles tendon contracture or equinovarus cavus deformity.
4. Signed informed consent form by patients/legal guardians for voluntary participation in the clinical study, with full comprehension of and commitment to study protocols .
5. Suboptimal response to standard conservative treatments (pharmacotherapy and/or rehabilitative exercise programs) with progressive worsening of gait abnormalities and foot deformities .
6. Functional impairment secondary to isolated Achilles tendon contracture or equinovarus cavus deformity, manifesting as ambulatory pain, frequent falls, and significant quality-of-life limitations.
7. Ability to ambulate barefoot for 10 meters independently or with assistive devices.

Exclusion Criteria:

1. Prior history of foot and ankle orthopedic surgery.
2. Severe cognitive impairment or an inability to adhere to postoperative protocols and functional assessments.
3. Isolated Achilles tendon contracture or equinovarus cavus deformity resulting from definitive etiologies (e.g., diabetes mellitus, infectious arthritis, or inflammatory arthropathy).
4. Significant peripheral vascular disease or clinically significant unstable medical conditions, including malignancies, hematologic disorders, and cardiopulmonary, hepatic, or renal insufficiency.
5. Coexisting neurodegenerative or neuromuscular disorders that are unrelated to hereditary spastic paraplegia (HSP).
6. Poor compliance with study requirements or other contraindications to participation in clinical trials.

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients meet the clinical and genetic diagnostic criteria of hereditary spastic paraplegia (HSP) between 10 to 45 years old with foot deformities.after undergoing standard conservative management (including pharmacological therapy and rehabilitation exercises) with suboptimal outcomes. Patients agree to participate in clinical trials and able to understand and comply with the research program.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society Score（AOFAS scores） | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  The quantitative assessment of ankle-foot function，directly reflects the long-term improvement in foot functionality following surgical intervention, serving as a critical indicator of therapeutic efficacy.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Score | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  The Visual Analog Scale (VAS) is a standardized tool for quantifying subjective symptoms (including pain and discomfort), serving as a critical indicator of surgical efficacy in alleviating foot pain in patients with Hereditary Spastic Paraplegia (HSP).
Foot Posture Index (FPI) | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  The Foot Posture Index (FPI) is a quantitative tool for assessing foot posture, designed to objectively evaluate the severity of foot alignment abnormalities.
6-Minute Walk Test (6MWT) | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  The 6-MWT measures the distance a person can walk in six minutes. A shorter distance indicates lower exercise capacity
Spastic Paraplegia Rating Scale (SPRS) | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  The change in the Spastic Paraplegia Rating Scale (SPRS) score : range: 0-52, higher scores mean a worse outcome
Gross Motor Function Measure-88 (GMFM-88) for Minors | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  Gross Motor Function Measure-88 (GMFM-88) score: range: 0-264, higher scores mean a better outcome

OTHER OUTCOMES:
MoCA score | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  Montreal Cognitive Assessment (MoCA) score: range: 0-30, higher scores mean a better outcome.
MMSE score | From the end of treatment to observations at 1 months, 3months, 6months, 12months, 18months, and 24months respectively.
  Mini-Mental State Examination (MMSE) : range: 0-30, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, phD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No